CLINICAL TRIAL: NCT04590105
Title: The Impact of a Smartphone App on the Quality of Pediatric Colonoscopy Preparations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, James Brief, Principal Investigator, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1132702
Record Dates: First submitted 2020-09-28; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Subjects were randomly assigned via block randomization to receive either written or software-based prep instructions.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Subjects were randomly assigned via block randomization to receive either written or software-based prep instructions. To eliminate bias, the four grading gastroenterologists who judged the quality of the subject's cleanout did not know whether subjects had used written or app instructions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App Subject (Experimental): Users who were assigned to use a smartphone app downloaded a free app from the iOS App or Google Play stores titled "SB Colonoscopy Prep." The app informed subjects about their colonoscopy procedure, alerts them when to take their medications throughout the hours-long colonoscopy prep process and tells them when to arrive to the endoscopy suite.
  Interventions: Device: Smartphone App "SB Colonoscopy Prep"
- Written Instruction Subjects (Active Comparator): Subjects in the control group were given a three-page document that described the procedure and instructed users on how to take the preparation medications. The written instructions had a list of frequently asked questions about colonoscopies and the URL of a website where users could view the animated video that was included in the app. The written instructions also contained the time and date of the procedure. All subjects were instructed to arrive one hour before their scheduled procedure.
  Interventions: Other: Written Instruction

INTERVENTIONS:
Device: Smartphone App "SB Colonoscopy Prep" — We created a smartphone app that informs patients about their colonoscopy procedure, alerts them when to take their medications throughout the hours-long colonoscopy prep process and tells them when to arrive to the endoscopy suite.
  Arms: App Subject
Other: Written Instruction — Written Instruction
  Arms: Written Instruction Subjects

SUMMARY:
The investigators developed a smartphone app that guides pediatric patients and their families through colonoscopy prep in an attempt to see if an app could improve the colonoscopy process.

DETAILED DESCRIPTION:
The investigators created a smartphone app designed for pediatric patients and their families that informs patients about their colonoscopy procedure, alerts them when to take their medications throughout the hours-long colonoscopy prep process and tells them when to arrive to the endoscopy suite. The investigators designed a study to determine if this app will yield improved colonoscopy cleanouts, better patient understanding of the procedure, fewer calls to the GI service and more punctual arrival times to the endoscopy suite compared to patients who receive written instructions that do not actively interact with the patient before, during or after their colonoscopy prep.

ELIGIBILITY:
Inclusion Criteria:

- Aged 5-18 years scheduled to undergo a diagnostic and/or therapeutic colonoscopy

Exclusion Criteria:

* Patients who had undergone a colonoscopy within the past one year
* Patients admitted for a nasogastric (NG) cleanout
* Patients requiring colonoscopy preparation medication other than Polyethylene Glycol
* Patients with poor understanding of English.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2014-11-15 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
Smartphone application use was associated with increased number of "excellent" colonoscopy preps. | Each subject was assessed from the time they were scheduled for their colonoscopy to the day of their procedure, up to three months for subjects. Subjects were scored on their colonoscopies immediately following the procedure once the patient was stable
  Prep quality was measured with the validated Boston Scoring Scale. A score of 0, 1, 2 or 3 is given to the right, transverse and left colon based on the amount and consistency of stool visualized as well as the ease or difficulty of guiding endoscopic instrumentation during a colonoscopy. Higher scores indicate a cleaner colon and as per Lai, a Boston Score of 7 or above indicates an "excellent" prep. To eliminate bias, the four grading gastroenterologists did not know whether subjects had used written or app instructions.

SECONDARY OUTCOMES:
The difference in the number of calls to the gastroenterology service between app users and controls. | Each subject was assessed from the time they were scheduled for their colonoscopy to the day of their procedure, up to three months for subjects
  Calls to the GI service were recorded by the GI staff.
The difference between app users and controls regarding patient arrival time. | Each subject was assessed from the time they were scheduled for their colonoscopy to the day of their procedure, up to three months for subjects
  Patient arrival time was taken from the patients arrival time in the endoscopy suite.
The significant difference between app users and controls regarding patient knowledge about the procedure. | Each subject was assessed from the time they were scheduled for their colonoscopy to the day of their procedure, up to three months for subjects
  A questionnaire with validated questions determined whether subjects improvement their knowledge before and after receiving colonoscopy information.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Morganstern, MD, Study Director — Stony Brook University Hospital

IPD SHARING:
Plan to Share IPD: Yes
I am happy to share all data in whatever way is easiest for everyone
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately
Access Criteria: Email request

REFERENCES:
- [Background] Pall H, Zacur GM, Kramer RE, Lirio RA, Manfredi M, Shah M, Stephen TC, Tucker N, Gibbons TE, Sahn B, McOmber M, Friedlander J, Quiros JA, Fishman DS, Mamula P. Bowel preparation for pediatric colonoscopy: report of the NASPGHAN endoscopy and procedures committee. J Pediatr Gastroenterol Nutr. 2014 Sep;59(3):409-16. doi: 10.1097/MPG.0000000000000447. PMID 24897169
- [Background] Pillai A, Menon R, Oustecky D, Ahmad A. Educational Colonoscopy Video Enhances Bowel Preparation Quality and Comprehension in an Inner City Population. J Clin Gastroenterol. 2018 Jul;52(6):515-518. doi: 10.1097/MCG.0000000000000893. PMID 28742732
- [Background] Hayat U, Lee PJ, Lopez R, Vargo JJ, Rizk MK. Online Educational Video Improves Bowel Preparation and Reduces the Need for Repeat Colonoscopy Within Three Years. Am J Med. 2016 Nov;129(11):1219.e1-1219.e9. doi: 10.1016/j.amjmed.2016.06.011. Epub 2016 Jul 6. PMID 27393880
- [Background] Park JS, Kim MS, Kim H, Kim SI, Shin CH, Lee HJ, Lee WS, Moon S. A randomized controlled trial of an educational video to improve quality of bowel preparation for colonoscopy. BMC Gastroenterol. 2016 Jun 17;16(1):64. doi: 10.1186/s12876-016-0476-6. PMID 27317249
- [Background] Lorenzo-Zuniga V, Moreno de Vega V, Marin I, Barbera M, Boix J. Improving the quality of colonoscopy bowel preparation using a smart phone application: a randomized trial. Dig Endosc. 2015 Jul;27(5):590-5. doi: 10.1111/den.12467. Epub 2015 Mar 20. PMID 25708251
- [Background] Kang X, Zhao L, Leung F, Luo H, Wang L, Wu J, Guo X, Wang X, Zhang L, Hui N, Tao Q, Jia H, Liu Z, Chen Z, Liu J, Wu K, Fan D, Pan Y, Guo X. Delivery of Instructions via Mobile Social Media App Increases Quality of Bowel Preparation. Clin Gastroenterol Hepatol. 2016 Mar;14(3):429-435.e3. doi: 10.1016/j.cgh.2015.09.038. Epub 2015 Oct 20. PMID 26492848
- [Background] Cook KA, Modena BD, Simon RA. Improvement in Asthma Control Using a Minimally Burdensome and Proactive Smartphone Application. J Allergy Clin Immunol Pract. 2016 Jul-Aug;4(4):730-737.e1. doi: 10.1016/j.jaip.2016.03.005. Epub 2016 Apr 20. PMID 27107690
- [Background] Iacoviello BM, Steinerman JR, Klein DB, Silver TL, Berger AG, Luo SX, Schork NJ. Clickotine, A Personalized Smartphone App for Smoking Cessation: Initial Evaluation. JMIR Mhealth Uhealth. 2017 Apr 25;5(4):e56. doi: 10.2196/mhealth.7226. PMID 28442453
- [Background] Voiosu A, Tantau A, Garbulet C, Tantau M, Mateescu B, Baicus C, Voiosu R, Voiosu T. Factors affecting colonoscopy comfort and compliance: a questionnaire based multicenter study. Rom J Intern Med. 2014;52(3):151-7. PMID 25509558
- [Background] Sagawa T, Sato K, Tomizawa T, Mizuide M, Yasuoka H, Shimoyama Y, Kuribayashi S, Kakizaki S, Kawamura O, Kusano M, Yamada M. A prospective randomized controlled trial of AJG522 versus standard PEG+E as bowel preparation for colonoscopy. Biomed Res Int. 2015;2015:521756. doi: 10.1155/2015/521756. Epub 2015 Jan 22. PMID 25688357
- [Background] Ting TV, Kudalkar D, Nelson S, Cortina S, Pendl J, Budhani S, Neville J, Taylor J, Huggins J, Drotar D, Brunner HI. Usefulness of cellular text messaging for improving adherence among adolescents and young adults with systemic lupus erythematosus. J Rheumatol. 2012 Jan;39(1):174-9. doi: 10.3899/jrheum.110771. Epub 2011 Nov 15. PMID 22089460
- [Background] Perski O, Blandford A, Ubhi HK, West R, Michie S. Smokers' and drinkers' choice of smartphone applications and expectations of engagement: a think aloud and interview study. BMC Med Inform Decis Mak. 2017 Feb 28;17(1):25. doi: 10.1186/s12911-017-0422-8. PMID 28241759
- [Background] Badawy SM, Kuhns LM. Economic Evaluation of Text-Messaging and Smartphone-Based Interventions to Improve Medication Adherence in Adolescents with Chronic Health Conditions: A Systematic Review. JMIR Mhealth Uhealth. 2016 Oct 25;4(4):e121. doi: 10.2196/mhealth.6425. PMID 27780795
- [Background] Iribarren SJ, Cato K, Falzon L, Stone PW. What is the economic evidence for mHealth? A systematic review of economic evaluations of mHealth solutions. PLoS One. 2017 Feb 2;12(2):e0170581. doi: 10.1371/journal.pone.0170581. eCollection 2017. PMID 28152012
- [Derived] Brief J, Chawla A, Lerner D, Vitola B, Woroniecki R, Morganstern J. The Impact of a Smartphone App on the Quality of Pediatric Colonoscopy Preparations: Randomized Controlled Trial. JMIR Pediatr Parent. 2020 Nov 10;3(2):e18174. doi: 10.2196/18174. PMID 33170131